CLINICAL TRIAL: NCT02343510
Title: Detection of Chlamydia DNA by Polymerase Chain Reaction ( PCR ) in Tumours Tissue of Primary Tubal and Ovarian Cancers : a Pilot Study
Brief Title: Detection of Chlamydia DNA by Polymerase Chain Reaction in Primary Tubal and Ovarian Cancers Tissues : a Pilot Study
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, dr mohamed laban, professor mohammed laban, Ain Shams University
Other Study IDs: lab7682
Record Dates: First submitted 2015-01-10; First posted 2015-01-22 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Malignant Neoplasm of Fallopian Tube
Keywords: Fallopian tubal cancer, high grade serous , ovarian cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Archival Paraffin blocks for cases of primary tubal cancers , high grade serous ovarian cancers , low grade serous ovarian cancers and normal Fallopian tubes removed during Hysterectomy operations for benign Gynecological indications
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- primary tubal cancer group: Paraffin blocks of cases of primary tubal cancer
  Interventions: Other: PCR for chlamydia DNA in primary tubal cancer
- high grade serous ovarian cancer group: Paraffin blocks of cases of high grade serous ovarian cancer
  Interventions: Other: PCR for chlamydia DNA in primary tubal cancer
- Low Grade Serous Ovarian Cancer: Paraffin blocks of cases of low grade serous ovarian cancer
  Interventions: Other: PCR for chlamydia DNA in primary tubal cancer
- normal tubes group: Paraffin blocks of tubes of hysterectomies due to non-oncologic causes
  Interventions: Other: PCR for chlamydia DNA in primary tubal cancer

INTERVENTIONS:
Other: PCR for chlamydia DNA in primary tubal cancer — PCR for presence of chlamydia DNA in paraffin blocks retrieved for tubal and ovarian tissues in all groups

SUMMARY:
PCR for chlamydia DNA is done in paraffin blocks of cases of primary tubal cancer and is compared to cases of high grade serous ovarian cancer and normal tubes .

DETAILED DESCRIPTION:
The investigators shall review the early cancer detection unite pathology records for the past 10 years , for cases diagnosed with primary Fallopian tube cancers , cases of high and low grade serous ovarian cancer and cases underwent hysterectomy and salpingectomy for non oncological reasons. Paraffin blocks for suitable selected patients will be examined histologically to confirm the primary diagnosis . Chlamydia DNA in these paraffin blocks of the Fallopian tubes and ovarian tissues will be examined using PCR techniques . The possible correlation between the presence of Chlamydia DNA and the ovarian serous tumours and primary tubal cancer will be analyzed statistically .

ELIGIBILITY:
Inclusion Criteria:

* any patient with primary tubal cancer and high grade serous cancer and normal tubes.

Exclusion Criteria:

* clinical pelvic inflammatory disease
* salpingectomy for ectopic

Ages: 40 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pathology blocks of patients with primary tubal cancer and with high grade serous ovarian cancer and normal tubes.
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2015-01; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Presence of chlamydia DNA in tubal and ovarian tissues | Up to 24 weeks

SECONDARY OUTCOMES:
Presence of concomitant tubal cancer with high grade serous ovarian cancer | Up to 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams Maternity Hospital, Cairo, Egypt